CLINICAL TRIAL: NCT01927185
Title: Long-versus Short-Axis Ultrasound Guidance for Subclavian Vein Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Vezzani Antonella, Chief of the Cardiac Surgery Intensive Care Unit, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16368
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Vascular Access Complication; Perioperative/Postoperative Complications
Keywords: central venous access; ultrasonography; subclavian vein; pneumothorax; vessel view
MeSH Terms: conditions — Postoperative Complications; Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long Axis strategy (Active Comparator): The central venous catheterization will be performed by the long axis approach
  Interventions: Device: Long Axis strategy
- Short Axis Strategy (Active Comparator): The central venous catheterization will be performed by the short axis approach
  Interventions: Device: Short Axis Strategy

INTERVENTIONS:
Device: Long Axis strategy — With the long-axis approach the vein appeared in the longitudinal view. With this approach only the vein was visible on the screen. The needle was held at a 30° angle, oriented in-plane with the transducer and the skin punctured at the base of the transducer. The vessel alignment was maintained during the procedure and the entire length of the needle was visible during the progression through the tissues.
  Arms: Long Axis strategy
Device: Short Axis Strategy — With the short-axis approach the probe was positioned almost perpendicularly to the clavicle. The needle was held at an angle of 45° relative to the skin surface and sagittal to the plane of the probe (out-of-plane). During the progression to the vessel, the visualization of the needle was limited to the deformation of tissue and artefacts produced by needle advancement. When the tip abutted the vein wall, additional pressure produced transient vessel deformation, which disappeared once the wall was penetrated.
  Arms: Short Axis Strategy

SUMMARY:
Central venous catheterization is commonly applied in patients undergoing cardiac surgery. The subclavian vein has lower risk of infection and provides more patients comfort. However central venous catheterization may results in complications such as pneumothorax, hemothorax or arterial puncture. It has been suggested that ultrasound (US) guidance could improve the success rate, reduce the number of needle passes and decrease complications. Two different real-time 2-dimensional US techniques can be employed in the insertion of central venous catheters. The first technique involves real-time US-guided cannulation of subclavian vein using a long axis/in-plane approach. The second one involves real-time US-guided using a short axis/out-off-plane approach. However to date no studies have compared their efficacy and safety. The purpose of this study was to compare the US-guided long-axis versus short-axis approach for the SCV catheterization in adult critical care patients.

DETAILED DESCRIPTION:
The two techniques used for vessel visualization are far different:

The Short-Axis (SA) approach attempts to view the vessel in cross-section while venous access is obtained. The strength of the SA approach is that the vein is centered under the transducer and that the midpoint of the transducer becomes a reference point for the insertion of the needle, and that at the same time is possible to visualize SC artery and the pleural line. SA approach is easy to learn by novice sonologists.

The Long-Axis (LA) approach employs a technique that views the length of the vessel during cannulation.For this reason, with LA approach is possible to visualize the needle advance during the entire procedure from the soft tissues until the lumen of the vein, but SC artery and pleural line are not visualized in the same scan. For LA approach, practice is required to keep the needle precisely within the image and care must be taken to avoid the probe inadvertently moving away from the target structure.

ELIGIBILITY:
Inclusion Criteria:

* aged =>18 years
* patients who needed central venous catheter for clinical reasons

Exclusion Criteria:

* aged <18a years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Success rate | up to 4 hours

SECONDARY OUTCOMES:
Access Time | Hours: 0,1
Central line-associated blood stream infection | days 0-21
Number of attempts | hours: 0-2
  Overall number of skin penetration and number of withdraws and redirections of the needle
Complication rate | Hours: 0-6-12-24
  Pneumothorax, Haemothorax, Hydrothorax, Artery puncture, Hematoma, Malpositions

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Vezzani, MD, Study Director — Cardiac Surgery. Azienda Ospedaliero Universitaria di Parma; Tiziano Gherli, MD, Study Chair — Cardiac Surgery. Azienda Ospedaliero Universitaria di Parma; Tullio Manca, MD, Principal Investigator — Cardiac Surgery. Azienda Ospedaliero Universitaria di Parma
Locations (1):
- Cardiac Surgery. Azienda Ospedaliero Universitaria di Parma, Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fragou M, Gravvanis A, Dimitriou V, Papalois A, Kouraklis G, Karabinis A, Saranteas T, Poularas J, Papanikolaou J, Davlouros P, Labropoulos N, Karakitsos D. Real-time ultrasound-guided subclavian vein cannulation versus the landmark method in critical care patients: a prospective randomized study. Crit Care Med. 2011 Jul;39(7):1607-12. doi: 10.1097/CCM.0b013e318218a1ae. PMID 21494105
- [Background] Matalon TA, Silver B. US guidance of interventional procedures. Radiology. 1990 Jan;174(1):43-7. doi: 10.1148/radiology.174.1.2403684.
- [Background] Abboud PA, Kendall JL. Ultrasound guidance for vascular access. Emerg Med Clin North Am. 2004 Aug;22(3):749-73. doi: 10.1016/j.emc.2004.04.003. PMID 15301849
- [Background] Blaivas M, Brannam L, Fernandez E. Short-axis versus long-axis approaches for teaching ultrasound-guided vascular access on a new inanimate model. Acad Emerg Med. 2003 Dec;10(12):1307-11. doi: 10.1111/j.1553-2712.2003.tb00002.x. PMID 14644780
- [Background] Blaivas M, Adhikari S. An unseen danger: frequency of posterior vessel wall penetration by needles during attempts to place internal jugular vein central catheters using ultrasound guidance. Crit Care Med. 2009 Aug;37(8):2345-9; quiz 2359. doi: 10.1097/CCM.0b013e3181a067d4. PMID 19531950
- [Background] Shah A, Smith A, Panchatsharam S. Ultrasound-guided subclavian venous catheterisation - is this the way forward? A narrative review. Int J Clin Pract. 2013 Aug;67(8):726-32. doi: 10.1111/ijcp.12146. PMID 23869675